CLINICAL TRIAL: NCT06019247
Title: Individual Placement and Support (IPS) for Serious Mental Illness in Jalisco, Mexico
Brief Title: Individual Placement and Support Mexico
Acronym: IPS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Collaborators: Instituto Jalisciense de Salud Mental (SALME) (Other); Research Foundation for Mental Hygiene, Inc. (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Ricardo Arturo Saracco Alvarez, UNDER DIRECTOR OF CLINICAL RESEARCH, Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IC22176.0
Record Dates: First submitted 2023-05-02; First posted 2023-08-31 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Severe Mental Disorder
Keywords: Individual placement and support; Serious mental illness; Jalisco; Mexico
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Our pilot RCT will examine both the implementation and effectiveness of IPS. We will use the Dynamic Adaptation Process model9 to adapt and implement IPS as well as to assess fidelity and identify barriers and facilitators. Then we will enroll 120 PSMI drawn from CAISAME-EP, which covers marginalized and poor communities. The outcomes of this pilot RCT will include employment, financial well-being, and health (i.e., symptoms and functioning). We will also quantify the cost of adapting and delivering IPS in this context. We will follow NIH guidelines on rigor and transparency to ensure strict application of the scientific method. Accordingly, we provide below detailed information regarding adaptation processes, recruitment, inclusion and exclusion criteria, outcomes and measures, and data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Services. (No Intervention): Generally, providers of rehabilitation Usual Care for PSMI at CAISAME-EP include 2 full-time psychologists, 2 full-time social workers, a half-time occupational therapist, and a half-time psychiatrist. This team, however, also provides services to clients with other mental conditions (e.g., substance use). As a result, the Usual Care services are of lower intensity than IPS and omit most of the key ingredients of the intervention. Moreover, it does not follow a standardized manual/protocol. The Usual Care team also offers other services such as psychiatric medication, individual and group psychotherapy, and psychoeducation for clients and relatives.
- Adapted IPS (Experimental): The IPS program adaptation process, will be conducted with 2 teams of providers, each consisting of an employment specialist, a case manager: psychologist, social worker and a psychiatrist, who will work in coordination to provide IPS services (each specialist will have between 15 and 20 clients). The IPS team will consist of providers and will be trained by the Research Adaptation Team in consultation and supervised. Weekly case-oriented supervision with a trained IPS supervisor, biweekly telephone contact, and telephone consultations as needed will help the IPS teams maintain high fidelity IPS. Following randomization, individuals assigned to receive IPS will be assigned to an IPS treatment team and will be introduced directly to their assigned case managers. Case management and IPS staff will be in close proximity to facilitate both IPS staff attendance at case management team meetings and the ongoing interaction necessary for efficient IPS implementation.
  Interventions: Other: Individual placement support (IPS)

INTERVENTIONS:
Other: Individual placement support (IPS) — IPS is the most studied psychiatric rehabilitation intervention in the world. It is based on eight principles: inclusion of all clients who have declared a desire to work, no pre-vocational training, benefits counseling, rapid job search, treatment team-level integration of vocational and clinical services, consideration of client preferences in all decisions, assistance in job development, provision of follow-up supports after finding employment, and a focus on competitive employment. We propose to adapt and pilot the IPS to improve employment and health among people with severe mental disorders in Mexico.
  Arms: Adapted IPS

SUMMARY:
There is substantial data to suggest that the Individual Placement and Support (IPS) model, a the investigatorsll-known, evidence-based practice, can help people with mental illness (PSMI) succeed in competitive employment (i.e., on average 55%, but over 60% in credible studies). Hothe investigatorsver, not a single country in Latin America offers IPS services. In addition, services to support employment and education tend to be ad hoc, low-intensity, and not the investigatorsll evaluated because most clinicians are not trained in evidence-based practices.

Clinicians are not trained in evidence-based approaches and do not provide high-fidelity services. The overall goal of this project is to pilot the IPS for PSMI in the Center for Comprehensive Care in Long-Stay Mental Health (CAISAME-EB, in Spanish), the largest mental health clinic in Jalisco, Mexico. CAISAME-EB integrates primary care and provides medication and psychosocial rehabilitation services to a large population of PSMI (n=~5,000). This team serves marginalized communities similar to other urban areas in low- and middle-income countries (LMICs) in Latin America and elsewhere.

The investigators will use the Dynamic Adaptation Process model to first inform the adaptation of IPS in Mexico, using our previous experience adapting IPS and deep understanding of the local context (e.g., the nature of the labor market in Mexico) to inform the adaptations. The investigators will then evaluate the implementation and impact of the adapted IPS in a pilot RCT (N = 120).

This pilot RCT will Include quantitative and qualitative assessments at baseline, 6 months, and 12 months with clients, providers, and other key stakeholders. The investigators aim to refine implementation processes, understand outcomes and tools, and estimate pothe investigatorsr for a future regional trial in Latin America.

DETAILED DESCRIPTION:
The researchers propose to adapt, implement, and evaluate the Individual Placement and Support (IPS) model for people with serious mental illness (PSMI) in Jalisco, Mexico. Substantial data indicate that IPS can help PSMI succeed in competitive employment (i.e., 55% on average, but over 60% in credible studies). In addition, successful employment through IPS has been shown to improve quality of life, self-esteem, and community integration, and to reduce symptoms, hospitalizations, and mental health costs. With the partial exception of Chile, no country in Latin America offers IPS services. Previous regional research has reported that PSMI experience extreme poverty, exclusion from educational and employment opportunities, and multiple traumas, including violence and abuse. Evidence-based, locally adapted initiatives to improve the living conditions and social inclusion of this vulnerable population are warranted.

In Mexico, mental health care for PSMI is often fragmented and does not follow evidence-based practices (EBP). The Jalisco Mental Health System, a large network of mental health facilities throughout the state of Jalisco, is an exception. The researchers plan to implement IPS at the Center for Comprehensive Care in Long-Stay Mental Health (CAISAME-EB, in Spanish), the largest mental health clinic in Jalisco. CAISAME-EB integrates primary care and provides medication and psychosocial rehabilitation services to a large population of PSMI (n=~5,000). The usual care services are of lower intensity than IPS and lack most of its key components.

This team serves marginalized communities similar to other urban areas in low- and middle-income countries (LMICs) in Latin America and elsewhere. In addition, the regional government of Jalisco has committed to expanding the implementation of the adapted IPS program if the trial is successful.

Ricardo Saracco (National Institute of Psychiatry Ramón de la Fuente Muñiz, INPRF) and Alejandro Aldana (Jalisco Institute of Mental Health, IJSM) have brought together key stakeholders to collaborate with researchers in the US (Susser, Dixon, Bello, Mascayano). All have extensive expertise in psychosis research and in the implementation of evidence-based mental health practices in a variety of contexts, including Latin America. In addition, the INPRF and IJSM teams have a long-standing relationship in Mexico and have recently collaborated with the US team on a study of the impact of the COVID-19 pandemic on health care workers (e.g., the Health Care Workers HEROES study).

The investigators will initially use the Dynamic Adaptation Process model9 to inform the adaptation of IPS in Mexico. The investigators note that IPS has been adapted for successful implementation in more than 20 countries and for marginalized communities within the US (e.g., Latinxs). This prior experience and our deep understanding of the local context (e.g., the nature of the nature of the labor market in Mexico) will inform the adaptations. Second, the researchers will evaluate the implementation and impact of the revised intervention in a pilot RCT (N = 120). This pilot RCT will include quantitative and qualitative assessments at baseline, 6, and 12 months, conducted with clients (e.g., employment, financial well-being of the investigators), providers (e.g., attitudes toward the intervention), and providers (e.g., attitudes toward the intervention), (e.g., attitudes toward EBP), and other key stakeholders (e.g., potential employers). The researchers primary goals are to refine implementation processes, understand outcomes and tools, and assess investigators for a future, regional trial in Latin America.

The investigators are already part of a network of investigators in Latin America resulting from a previous NIMH grant (i.e., "RedeAmericas", contact PI Susser) that includes many investigators who would be willing and able to conduct a regional trial.

ELIGIBILITY:
Inclusion Criteria (Potential participants will be deemed eligible if they)

* Meet requirements for PSMI.
* Are receiving services from CAISAME-EP for at least one month.
* Are at least 18 years old.
* Have expressed a goal of paid, competitive employment.
* Have attended 2 informational sessions prior to recruitment.
* Have no competitive employment during the past 3 months.
* Are physically and cognitively able to participate in study for the planned year of follow-up.
* Are willing to provide informed consent.
* Agree not to seek usual vocational services.

Exclusion Criteria (Potential participants will not be eligible if they)

* Don't meet requirements for PSMI.
* Are not receiving services from CAISAME-EP for at least one month.
* Are not at least 18 years old or older than 60 years old.
* Have not expressed a goal of paid, competitive employment.
* Have not attended 2 informational sessions prior to recruitment.
* Have a competitive employment during the past 3 months.
* Are not physically and cognitively able to participate in study for the planned year of follow-up.
* Are not willing to provide informed consent.
* Don't agree not to seek usual vocational services.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
IPS Employment impact measure | One year
  The aim of the evaluation is to measure the impact of the IPS programme on the employability of the participants. Outcome measures will be based on a baseline interview and quarterly interviews with participants. The impact of the intervention will be measured by changes from baseline in time in jobs held, hours worked and wages earned.
Assessment of psychiatric symptoms | One year
  Indicators of participants' mental well-being will be measured at baseline, six months and twelve months. Psychiatric symptoms will be measured using the Colorado Symptom Index.
Assessment of mental and physical functioning. | One year
  Outcomes of physical and mental functioning in daily life will be measured at baseline, six months and twelve months using the Study Short-Form 12-Item and physical and mental functioning at work using the Functional Assessment Battery.

SECONDARY OUTCOMES:
Baseline customer demographics. | six months
  Participants will be interviewed at baseline prior to randomisation. Outcome demographic data will include age, ethnicity, gender, educational attainment, marital status, employment and financial status. Additional data will describe housing, justice system involvement, social capital and health service use.
Quarterly client employment interviews | six months
  Quarterly client interviews will document past-quarter employment, including jobs held, hours worked, and wages earned. Interviews will document job termination during quarters when jobs ended. The interviews will take place at CAISAME-EP if/when possible, considering the constraints imposed by the COVID-19 pandemic. When clients are unavailable for interview, a research assistant in Mexico will make several efforts to track and schedule the interview until the next interview period. Next interviews can track employment during missed intervals. These delays do not typically compromise data quality because the data describe continuous data collapsed over specified periods.
Follow-up interviews. | one year
  The follow-up interviews, conducted at 6 and 12 months after randomisation, complement the quarterly employment interview and include measures of health and functioning that mirror those administered at baseline. Additional data will be collected on housing, social capital and health service use. The follow-up interviews are conducted at the same time as the corresponding quarterly employment interviews. As with the quarterly employment interviews, if clients are unavailable for the follow-up interview, the research assistant will make several efforts to track and schedule the interview until the next quarterly interview period.
IPS Participation Measure | one year
  Monthly client interviews document the employment specialist's engagement with participants and the number of times and length of contact with the participant in job search activities. The type and number of job search activities in which participants have been involved are also recorded in the interview.
Employment specialist service log (time spent direct services, collaborating with mental health experts and job support). | six months
  Once a month, employment specialists complete service logs describing IPS service provision over the past week. Collecting this data on a time-sampling basis has been shown to be more reliable than using a continuous measure. Specialist activities documented will include time spent providing both direct (vs indirect) and community (vs office) services, as well as time spent working with mental health clinicians in the clinic, working on job development, and working on job support. These times can be compared to current IPS programme standards associated with high fidelity and assessed in relation to the adaptations resulting from the Dynamic Adaptation Process.
Participant employment report (weeks worked, hours worked per week, hourly wage, start and end dates of work) and feedback to IPS teams. | Eighteen months
  Quarterly client interviews will report on employment in the previous quarter, including jobs held, hours worked and wages earned. Interviews will document job quits in quarters in which jobs ended. If clients are unavailable for interview, a research assistant in Mexico will make several efforts to track and schedule the interview until the next interview period. Subsequent interviews may document employment during missed intervals. These delays do not usually affect the quality of the data, as the data describe continuous data that are aggregated over specific time periods.
  Summaries of the Employment Specialist's reports are provided to the IPS Team Leaders to monitor implementation and address potential issues in collaboration with the IPS teams and IPS TA/QA.

CONTACTS AND LOCATIONS:
Overall Officials: JESUS A. ALDANA LOPEZ, MPH, Study Chair — Jalisco Institute of Mental Health (SALME)
Locations (3):
- United States (2):
  - Columbia University, New York, New York
  - Research Foundation of Mental Hygiene, New York, New York
- Instituto Jalisciense de Salud Mental, Zapopan, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No